CLINICAL TRIAL: NCT04773249
Title: Comparison of Clinical and Ultrasonographic Efficacy of Two Different Splints Used in the Treatment of Lateral Epicondylitis: A Prospective Randomized Controlled Study
Brief Title: Comparison of Two Different Splints in the Treatment of Lateral Epicondylitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Banu Dilek, Assoc Prof, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DokuzEUKadir
Record Dates: First submitted 2021-02-21; First posted 2021-02-26 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Lateral Epicondylitis; Tennis Elbow
Keywords: ultrasonography; lateral epicondylitis bandage; wrist extension splint; wait-and-see policy; orthotic devices; forearm braces
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator
Masking Description: Single (Clinician)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lateral Epicondylitis Bandage (Experimental): A lateral epicondylitis bandage will be given to the patient for 6 weeks. The bandage will be positioned 5 cm distal to the lateral epicondyle to allow for elbow flexion. After the application, patients will be asked to punch and the belt on the band will be tightened. After the patients are asked to open the fist, the suitability of the pressure applied to the forearm will be evaluated. Patients will be asked to repeat this application while wearing the band. The patients will also be asked to use the bandage throughout the day, and to remove them during bathing and sleeping.
  Interventions: Device: Lateral Epicondylitis Bandage
- Wrist Extension Splint (Experimental): A wrist extension splint will be given to the patient for 6 weeks. The splint will be used to keep the wrist at 15-20 degrees of extension and to wrap the distal wrist and forearm without hindering finger movements. The patients will be asked to use the splint throughout the day, and to remove them during bathing and sleeping.
  Interventions: Device: Wrist Extension Splint
- Wait-and-see Policy (No Intervention): These patients will be monitored with a wait-and-see policy. No splint or band will be given to the patient.

INTERVENTIONS:
Device: Lateral Epicondylitis Bandage — The lateral epicondylitis bandage was first used by Ilfeld in 1965, and it is a non-elastic band that prevents the expansion of the muscles in the proximal forearm. A lateral epicondylitis bandage will be given to the patient for 6 weeks. The bandage will be positioned 5 cm distal to the lateral epicondyle to allow for elbow flexion. After the application, patients will be asked to punch and the belt on the band will be tightened. After the patients are asked to open the fist, the suitability of the pressure applied to the forearm will be evaluated. Patients will be asked to repeat this application while wearing the band. The patients will also be asked to use the bandage throughout the day, and to remove them during bathing and sleeping.
  Other Names: Elbow Band; Counterforce Elbow Strap; Epicondylitis Bandage; Lateral Epicondyle Bandage
  Arms: Lateral Epicondylitis Bandage
Device: Wrist Extension Splint — Wrist extension splint is an upper extremity orthosis that keeps the wrist at 15-20 degrees of extension with the polyethylene bar it contains. A wrist extension splint will be given to the patient for 6 weeks. The splint will be used to keep the wrist at 15-20 degrees of extension and to wrap the distal wrist and forearm without hindering finger movements. The patients will be asked to use the splint throughout the day, and to remove them during bathing and sleeping.
  Other Names: Hand-wrist Resting Orthosis; Wrist Splint
  Arms: Wrist Extension Splint

SUMMARY:
Lateral epicondylitis (LE) or tennis elbow; is the most common cause of lateral pain in the elbow, with an incidence of 1-3% in the general population. It is thought to develop as a result of overuse inflammation of the wrist joint extensor tendons, originating from the lateral epicondyle of the humerus. The most common symptom is the pain located in the lateral aspect of the elbow, which can spread across the forearm extensor face and is aggravated by wrist extension, forearm supination, and strong grip movements of the hand. The diagnosis is made by clinical and ultrasonographic evaluations. Significant correlations were found between clinical symptoms of LE and increased joint extensor tendon thickness, focal hypoechogenicity, intratendinous calcification, bone abnormality, and diffuse heterogeneity findings that can be monitored by diagnostic ultrasound. Wait-see policy, conservative treatment regimens, local injections, and surgical approaches are the treatment methods that can be used on a patient-based basis until today. Conservative treatment options include physical therapy modalities such as exercise, massage, laser, electrotherapy, therapeutic ultrasound, extracorporeal shock wave therapy, the use of various splints, ice application, activity modification, rest, NSAIDs, and taping methods. The two prominent bracing methods are the lateral epicondylitis band and the wrist extension splint. Although these two methods are frequently used in daily practice, the limitations of studies investigating the effectiveness of orthoses and which orthosis are more effective draw attention. In comparative studies, some factors may affect clinical results such as allowing patients to use NSAIDs when necessary and organizing a home exercise program. Besides, none of them included a control group and the patients were not evaluated by ultrasonography. This study aims to compare the effects of the use of two different splints (lateral epicondylitis band and wrist extension splint) on clinical and ultrasonographic parameters in patients with a diagnosis of lateral epicondylitis.

DETAILED DESCRIPTION:
The study is randomized and controlled. 158 patients will be included in to study who apply to Dokuz Eylül University Faculty of Medicine, Department of Physical Medicine and Rehabilitation Clinic with the complaint of elbow pain, aged between 18-65 years and diagnosed with lateral epicondylitis by clinical and ultrasonographic methods. These patients will be divided into three groups randomly (group1 n:53, group 2 n:53, group 3 n:52).

First group: A lateral epicondylitis bandage will be given to the patient for 6 weeks. The bandage will be positioned 5 cm distal to the lateral epicondyle to allow for elbow flexion. After the application, patients will be asked to punch and the belt on the band will be tightened. After the patients are asked to open the fist, the suitability of the pressure applied to the forearm will be evaluated. Patients will also be asked to repeat this application while wearing the band.

Second group: A wrist extension splint will be given to the patient for 6 weeks. The splint will be used to keep the wrist at 15-20 degrees of extension and to wrap the distal wrist and forearm without hindering finger movements.

Third group: These patients will be monitored with a wait-and-see policy. No splint or band will be given to the patient.

Before treatment, age, gender, occupation, body mass index, duration of symptoms, trauma history, dominant hand, side of the symptom and previous similar complaint history will be questioned in all three groups.

All of the patients will be asked not to lift heavy for 6 weeks, to use their splints throughout the day, and to remove them during bathing and sleeping. Throughout the study, all patients will be allowed to take only paracetamol oral tablets as pain relief if needed and will be asked to keep a medication diary.

All patients will be evaluated 3 times, before the treatment, in the 3rd week during the treatment process, and in the 6th week after the treatment with a visual analog scale, patient-rated tennis elbow evaluation questionnaire, hand dynamometer, and ultrasonographic measurements. All evaluations will be done blindly by the clinician.

The primary aim of this randomized controlled single-blind study is to compare the effects of lateral epicondylitis bandage and wrist extension splint treatment on ultrasonographic changes in patients with lateral epicondylitis. Ultrasonographic evaluations will include measurement of maximum tendon thickness and assessment of hypoechogenicity, heterogeneity, neovascularity, and bone abnormality. The maximum tendon thickness in the capitellar and radiocapitellar regions of the common extensor tendon will be measured for both upper extremities.

The secondary aim is to compare the effects of these two different splint treatments on clinical changes such as pain, functional disability, sensitivity, and handgrip strength. Pain and functional disability will be measured by the Visual Analog Scale and Patient Rated Tennis Elbow Evaluation questionnaire, the sensitivity will be measured by algometer, and handgrip strength will be measured by hydraulic hand dynamometer for both hands.

ELIGIBILITY:
Inclusion Criteria:

* Applying to Dokuz Eylül University Medical Faculty Physical Medicine and Rehabilitation Department outpatient clinic
* Having pain in the elbow for less than 12 weeks and having no similar attack history for 1 year
* Diagnosing lateral epicondylitis with clinical and ultrasonographic evaluation
* Having pain of at least 3 in their VAS scores
* Agreeing to participate in the study

Exclusion Criteria:

* Having elbow pain for more than 12 weeks
* Having signs of lateral epicondylitis in the other extremity
* Having a history of injection for lateral epicondylitis
* In the last 3 months, who had physical therapy for lateral epicondylitis
* Having a history of elbow surgery and fracture in the elbow area.
* Having muscle weakness in the upper extremity due to cervical radiculopathy and/or entrapment neuropathy
* Having malignancy or neurological, rheumatological, and psychiatric disease comorbidities
* Pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-09-06 (Estimated)

PRIMARY OUTCOMES:
Change of the maximum tendon thickness of the common extensor tendon via ultrasonographic measurement | All patients will be evaluated 3 times, before treatment, third week of the treatment, and sixth week of the treatment with ultrasonographic measurements.
  The maximum tendon thickness in the capitellar and radiocapitellar regions of the common extensor tendon
Change of the hypoechogenicity of the common extensor tendon via ultrasonographic assessment. | All patients will be evaluated 3 times, before treatment, third week of the treatment, and sixth week of the treatment with ultrasonographic assessments.
  The assessment of hypoechogenicity of the common extensor tendon, Grade 0: Normal fibrillar and hypoechoic structure, Grade 1: hypoechoic lesions affecting less than 30% of whole section of the tendon, Grade 2: hypoechoic lesions affecting more than 30% and less than 50% of the whole section of the tendon, Grade 3: single large or multiple hypoechoic lesions affecting more than 50% of the whole section of the tendon / high-grade tendinosis.
Change of the heterogeneity of the common extensor tendon via ultrasonographic assessment. | All patients will be evaluated 3 times, before treatment, third week of the treatment, and sixth week of the treatment with ultrasonographic assessments.
  The assessment of heterogeneity of the common extensor tendon, Grade 1 = presence, Grade 0 = absence
Change of the neovascularity of the common extensor tendon via ultrasonographic assessment. | All patients will be evaluated 3 times, before treatment, third week of the treatment, and sixth week of the treatment with ultrasonographic assessments.
  The assessment of neovascularity of the common extensor tendon, Grade 0 = no detectable neovessels Grade 1 = neovessels detected in less than 30% of the whole section of the tendon Grade 2 = neovessels detected in more than 30% but less than 50% of the whole section of the tendon Grade 3 = neovessels detected in more than 50% of the whole section of the tendon.
Change of the bone abnormality of the lateral epicondyle via ultrasonographic assessment | All patients will be evaluated 3 times, before treatment, third week of the treatment, and sixth week( of the treatment with ultrasonographic assessments.
  The assessment of bone abnormality of the lateral epicondyle, Grade 1 = presence, Grade 0 = absence

SECONDARY OUTCOMES:
Change of the pain on the lateral elbow via Visual Analog Scale | All patients will be evaluated 3 times, before treatment, third week of the treatment, and sixth week of the treatment.
  The pain during rest, night, and daily life activities will be measured with a Visual Analog Scale (Minimum value : 0 , Maximum value: 100, A higher score indicates greater pain intensity.)
Change of the pain on the lateral elbow via Patient Rated Tennis Elbow Evaluation | All patients will be evaluated 3 times, before treatment, third week of the treatment, and sixth week of the treatment.
  The pain will be also measured by the Patient Rated Tennis Elbow Evaluation questionnaire.(which describe the pain on a scale from 0 to 10 for each of the 5 different questions. A higher score indicates greater pain intensity.)
Change of the functional disability via Patient Rated Tennis Elbow Evaluation | All patients will be evaluated 3 times, before treatment, third week of the treatment, and sixth week of the treatment.
  Functional disability will be measured by the Patient Rated Tennis Elbow Evaluation questionnaire. ( The best value = 0 , the worst value = 50.)
Change of the sensitivity via algometer | All patients will be evaluated 3 times, before treatment, third week of the treatment, and sixth week of the treatment.
  Sensitivity will be measured by an algometer as the value at which the pain first appears.
Change of the handgrip strength via hand dynamometer | All patients will be evaluated 3 times, before treatment, third week of the treatment, and sixth week of the treatment.
  Handgrip strength will be measured by a hydraulic hand dynamometer. Average values will be determined by making 3 separate measurements for both hands, and 30-second rest periods will be given between measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Banu Dilek, Assoc Prof, Study Chair — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Songur K, Demir ZD, Baysan C, Dilek B. Clinical and Ultrasonographic Effectiveness of Two Different Splints Used for the Treatment of Lateral Epicondylitis: A Prospective Randomized Controlled Study. Arch Phys Med Rehabil. 2024 Apr;105(4):655-663. doi: 10.1016/j.apmr.2023.12.010. Epub 2023 Dec 30. PMID 38163530